CLINICAL TRIAL: NCT01431378
Title: Pilot Study of Model Based Iterative Reconstruction Using 64-Slice Multidetector-Row CT Datasets Obtained From the Central Nervous System, Thorax, and Abdomen
Brief Title: Pilot Study of Model Based Iterative Reconstruction Using 64-Slice
Acronym: MBIR
Status: Terminated | Type: Observational
Why Stopped: Feasibility study, sufficient amount of data collected.
Sponsor: GE Healthcare (Industry)
Collaborators: American College of Radiology - Image Metrix (Industry)
Responsible Party: Sponsor
Other Study IDs: 106-2010-GES-0010
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Posterior Fossa Hemorrhage; Lung Cancer; Flank Pain; Urolithiasis; Focal Hepatic Necrosis
Keywords: CT scan; CNS; Thorax; Abdomen; staging of a known or suspected lung cancer; suspected urolithiasis; known or suspected focal liver lesion
MeSH Terms: conditions — Intracranial Hemorrhages; Lung Neoplasms; Flank Pain; Urolithiasis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CNS: CNS: Known or suspected pathology in the posterior fossa
- Thorax: Thorax: Patients referred for staging of a known or suspected lung cancer
- Abdomen 1: Abdomen: Patients with acute flank pain and suspected urolithiasis
- Abdomen 2: Abdomen: Patients with a known or suspected focal liver lesion

SUMMARY:
This study is being performed to confirm that the new technique, Model-Based Iterative Reconstruction (MBIR) with reduced radiation dose can deliver equivalent image quality for CT scans compared to current techniques (Filtered Back Projection with Adaptive Statistical Iterative Reconstruction (FBP with ASiR) and also to demonstrate that MBIR can improve general image quality characteristics at equivalent radiation dose levels.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Men or Women 30 years of age or older voluntarily willing to sign an informed consent.
* Patients indicated for one of the following:

CNS: Known or suspected pathology in the posterior fossa Thorax: Patients referred for staging of a known or suspected lung cancer Abdomen: Patients with acute flank pain and suspected urolithiasis or Abdomen: Patients with a known or suspected focal liver lesion

Exclusion Criteria:

* Subjects less than 30 years of age
* Pregnant women as confirmed by urine test or current accepted institution standard
* If IV contrast is required:
* Severe or uncontrolled allergy to iodinated contrast media
* Serum creatinine > 1.7 mg/dl or estimated glomerular filtration rate [eGFR] of <60 mg/min as recorded in medical file or by current accepted institution standard
* Unable or unwilling to provide written informed consent by self or legal guardian at the time of study enrollment
* Unstable physical condition as identified by physician

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population to include women or men 30 years of age or older referred for a CT scan
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Evidence for reduced x-ray radiation exposure for applicable patient indications | Side by side comparison once both scans have been performed
  Ultra-low radiation dose images reconstructed with MBIR yield similar anatomic and pathologic information compared to routine radiation dose images reconstructed with Filtered Back Projection (FBP) in the central nervous system (CNS), thorax, and abdomen.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Froedtert Memorial Lutheran Hospital, Miwaukee, Wisconsin